CLINICAL TRIAL: NCT04372901
Title: Passive Fit of CAD/CAM Implant Supported Screw-retained Metal Frameworks Based on Actual Versus Screwmented Ones Based on Virtual Implant Position: A Randomized Clinical Trial
Brief Title: Passive Fit of CAD/CAM Screw-retained Metal Frameworks Versus Screwmented Ones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed El-Sayed Mohamed Kamel, Master student- Oral implantology -Cairo univeristy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123987
Record Dates: First submitted 2020-04-24; First posted 2020-05-04 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Edentulous; Jaw
Keywords: Passive; Fit; Screwmented; CAD/CAM; Frameworks
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Intervention Model Description: Trial design to be conducted is RCT, split mouth , two arms, and Equivalence frame with 1:1 allocation ratio.
Masking Description: The study is based on different technical procedures of fabrication of the frameworks. Since these differences are visible, the operator, the assessor and the technician involved in the study cannot be blinded. Since blinding was not possible, randomization was delayed till the prosthetic phase to avoid any performance bias in the surgical steps. But the statistician will be blinded .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digitally constructed frameworks before implant placement (Experimental): Intervention group in which the edentulous area will be restored with 3-implant screwmented CAD/CAM frameworks constructed based on planned implant positions.
  Interventions: Procedure: Digitally constructed frameworks before implant placement
- digitally constructed frameworks after implant placement (Active Comparator): Control group: edentulous area will be restored with 3-implant conventional screw retained CAD/CAM frameworks constructed after implant placement
  Interventions: Procedure: Digitally constructed frameworks after implant placement

INTERVENTIONS:
Procedure: Digitally constructed frameworks before implant placement — Intervention group in which the edentulous area will be restored with 3-implant screwmented CAD/CAM frameworks constructed based on planned implant positions.
  Arms: digitally constructed frameworks before implant placement
Procedure: Digitally constructed frameworks after implant placement — Control group: edentulous area will be restored with 3-implant conventional screw retained CAD/CAM frameworks constructed after implant placement.
  Arms: digitally constructed frameworks after implant placement

SUMMARY:
CAD/CAM (computer aided design/ computer aided manufacturing) constructed screw retained implant supported frameworks give solutions for the problems arising from the lost wax technique by improving accuracy, adaptation and passive fit of the final restoration. However, concerns about the passive fit of a pre-implant insertion CAD/CAM constructed framework still exists due to the expected errors in imaging, registration, surgical guide construction, adaptation and hence transferring the planned position intra-orally.

DETAILED DESCRIPTION:
9. PICO Format: Population: mandibular free end saddle requiring 2 implants. Intervention: Digitally fabricated screw-mented retained metal frameworks constructed before implant placement Control: Digitally fabricated screw retained metal frameworks constructed after implant placement

Outcome:

Outcome Measuring device Measuring unit Passive fit One screw test Binary 13 Screw resistance Binary Radiographic ( digital periapical radiography) Binary III. Methods A) Participants, interventions & outcomes 9. Study settings: i. The study will be conducted at Department of Oral Implantology, faculty of oral and dental medicine, Cairo University, Egypt. ii. Participants will be selected from the outpatient clinic of implantology department, faculty of oral and dental medicine, Cairo University, Egypt. 10. Eligibility criteria: A-Inclusion criteria: i- Mandibular Kenndy Class I. ii- Opposing completely dentulous, fully or partially restored dentition. iii- Good oral hygiene. iv- The patient should have bone for implants, minimum bone height 10 mm and minimum bone diameter should be 6 mm. v- Adequate inter arch space for restoration 15mm or more. vi- Adult patients age ≥18 years B- Exclusion criteria: i. any medical disorder that could complicate surgical phase or affect osteointegration. Radiation chemotherapy. ii. smokers more than 10/daily. iii. Uncooperative patients. iv. Patients with Para-functional habits v. Patients with severe periodontal diseases. vi. Patients with limited mouth opening. vii. Presence of intraoral pathological lesions. viii. Diabetic (HbA1c >7.5%).

ELIGIBILITY:
.Inclusion Criteria:

* Mandibular Kenndy Class I.
* Opposing completely dentulous, fully or partially restored dentition.
* Good oral hygiene.
* The patient should have bone for implants, minimum bone height 10 mm and minimum bone diameter should be 6 mm.
* Adequate inter arch space for restoration 15 mm or more.
* Adult patients age ≥18 years

Exclusion Criteria:

* - . any medical disorder that could complicate surgical phase or affect osteointegration. Radiation chemotherapy.
* ii. smokers more than 10/daily.
* iii. Uncooperative patients.
* iv. Patients with Para-functional habits
* v. Patients with severe periodontal diseases.
* vi. Patients with limited mouth opening.
* vii. Presence of intraoral pathological lesions.
* viii. Diabetic (HbA1c >7.5%)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Passive fit | 10 weeks
  Evaluation of Passive fit between CAD/CAM Implant Supported Screw-retained Metal Frameworks Based on Actual Versus Screwmented Ones Based on Virtual Implant Position using one screw test .

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El-Sayyed, BDS, Principal Investigator — Teaching assistant MIU; Mohamed ElKhashab, Phd, Study Director — Lecturer of prosthodontics, Faculty of Dentistry, Cairo Univerusty; Iman Radi, Phd, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
The author of "study will publish it in an internationally acknowledged journal.

REFERENCES:
- [Background] de Franca DG, Morais MH, das Neves FD, Barbosa GA. Influence of CAD/CAM on the fit accuracy of implant-supported zirconia and cobalt-chromium fixed dental prostheses. J Prosthet Dent. 2015 Jan;113(1):22-8. doi: 10.1016/j.prosdent.2014.07.010. Epub 2014 Sep 30. PMID 25277028